CLINICAL TRIAL: NCT02044302
Title: A Prospective Randomized Double Blind Trial to Reduce Post-Operative Pain in Implant Based Breast Reconstruction
Brief Title: A Prospective Trial to Reduce Post-Operative Pain in Implant Based Breast Reconstruction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1304011938
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Post-operative Pain
Keywords: pain; breast cancer; breast implant; breast reconstruction
MeSH Terms: conditions — Pain, Postoperative; Pain; Breast Neoplasms | interventions — Bupivacaine; Botulinum Toxins; Botulinum Toxins, Type A; Analgesics; Narcotics; Morphine; Hypnotics and Sedatives; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- standard analgesics (Active Comparator): Current standard post-operative care for expander-implant breast reconstruction surgery consists of conventional pain medications including narcotics (like morphine, etc.) and sedatives (like valium). Placebo application during surgery will be made to establish perfection in the study design in terms of randomization and blinding. Injections will be done intramuscularly to the main chest muscle (pectoralis major) by the surgeon.
  Interventions: Drug: Analgesics
- standard analgesics and bupivacaine (Experimental): Current standard post-operative care for expander-implant breast reconstruction surgery consists of conventional pain medications including narcotics (like morphine, etc.) and sedatives (like valium). Patients will receive through an injection into the chest 10 ml (about 2 teaspoons) of 0.5% bupivacaine during surgery. Injections will be done intramuscularly to the main chest muscle (pectoralis major) by the surgeon.
  Interventions: Drug: Bupivacaine; Drug: Analgesics
- standard analgesics and botulinum toxins (Experimental): Current standard post-operative care for expander-implant breast reconstruction surgery consists of conventional pain medications including narcotics (like morphine, etc.) and sedatives (like valium). Patients will receive through an injection into your chest 50 U of Botox diluted in 4ml (about 1 teaspoon) of normal saline per breast during your operation. Injections will be done intramuscularly to the main chest muscle (pectoralis major) by the surgeon.
  Interventions: Drug: Botulinum Toxins; Drug: Analgesics
- standard analgesics, bupivacaine and botulinum toxins (Experimental): Current standard post-operative care for expander-implant breast reconstruction surgery consists of conventional pain medications including narcotics (like morphine, etc.) and sedatives (like valium). Patients will receive through an injection into your chest 10 ml (about 2 teaspoons) of 0.5% bupivacaine and 50 U of Botox diluted in 4ml (about 1 teaspoon) of normal saline per breast during the operation. Injections will be done intramuscularly to the main chest muscle (pectoralis major) by the surgeon.
  Interventions: Drug: Bupivacaine; Drug: Botulinum Toxins; Drug: Analgesics

INTERVENTIONS:
Drug: Bupivacaine
  Other Names: Exparel; Marcaine; Sensorcaine
  Arms: standard analgesics and bupivacaine; standard analgesics, bupivacaine and botulinum toxins
Drug: Botulinum Toxins
  Other Names: Botox
  Arms: standard analgesics and botulinum toxins; standard analgesics, bupivacaine and botulinum toxins
Drug: Analgesics
  Other Names: narcotic; morphine; sedative; valium

SUMMARY:
The investigators hypothesize that in mastectomy patients with breast reconstruction, the addition of bupivacaine and botulinum toxin (BT) will result in better pain control in the acute and chronic setting, compared to traditional pain management techniques which rely almost exclusively on opioid analgesics and sedatives like diazepam (valium). This expectation is based on the fact that bupivacaine produces pre-emptive analgesia and BT will produce muscle relaxation, the combination of which will target different sites of pain generation, thus producing better analgesia. We also hypothesize that additional benefits may accrue from this regimen including decreased nausea and vomiting, sedation and constipation as a result of diminished opioid use1.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing immediate unilateral or bilateral tissue expander breast reconstruction following therapeutic skin-sparing or nipple-sparing mastectomy requiring postoperative expansions
* Women undergoing immediate bilateral tissue expanders breast reconstruction following risk-reduction (prophylactic) skin-sparing or nipple-sparing mastectomy requiring postoperative tissue expansions.

Exclusion Criteria:

* Subjects who are unable to read or speak English;
* Breast reconstruction using the latissimus dorsi flap combined with a tissue expander;
* Documented diagnosis of chronic pain, chronic migraine, upper limb spasticity, cervical dystonia, axillary hyperhidrosis, strabismus or blepharospasm;
* Hypersensitivity to any botulinum toxin (BT) preparation or to any of the components in the formulation;
* Infection at the proposed site of injection;
* Pre-existing neuromuscular disorders (including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis);
* Aminoglycosides intake at the time of surgery (these antibiotics can potentiate the effect of BT);
* Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kwei, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blinded Group A | Blinded Group B
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — study terminated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Only two subjects were enrolled into 1 of the 2 blinded arms and then the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Group A | Blinded Group B | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Questionnaire
Description: The patient records their feeling of pain scaled in a subjective scale from 0 to 10. 0 means that there is no pain and 10 means that the worst pain you had. The other numbers mean that pain is in perceived as in between. The investigator will also mark a pain score in the facial expression scale of Mosby© by evaluating your facial appearance.
Time Frame: Post Operation Day 1
Population: The study was terminated after 2 subjects enrolled and outcomes were never fully collected not summarized.
Arm/Group | Terminated Cohort
Number analyzed (Participants) | 0

2. Secondary Outcome: Pain Score Questionnaire
Description: The patient records their feeling of pain scaled in a subjective scale from 0 to 10. 0 means that there is no pain and 10 means that the worst pain. The other numbers mean that pain is perceived as in between. The investigator will also mark a pain score in the facial expression scale of Mosby© by evaluating your facial appearance.
Time Frame: Post Operation Week 1
Population: The study was terminated after 2 subjects enrolled and outcomes were never summarized.
Arm/Group | Terminated Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Score Questionnaire
Description: as for outcome 2
Time Frame: Post Operation One Month
Population: The study was terminated after 2 subjects enrolled and outcomes were never summarized.
Arm/Group | Terminated Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Terminated Cohort
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes